CLINICAL TRIAL: NCT07339618
Title: Effects of Non-pharmacological Auditory and Somatosensory Stimulation on the Efficiency and Quality of Emergence From General Anesthesia
Brief Title: Non-pharmacological Auditory and Somatosensory Stimulation in Anesthetic Emergence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Guizhi Du, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChinaHospital 2025（1900）
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: General Anesthetic; Electroencephalographic
Keywords: General anesthesia; Emergence; Verbal stimulation; Somatosensory stimulation; EEG; Recovery of consciousness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Verbal Stimulation Group: (Active Comparator)
  Interventions: Behavioral: Verbal Stimulation
- Shoulder Tapping Group (Experimental)
  Interventions: Behavioral: Shoulder Tapping
- Shoulder Shaking Group (Experimental)
  Interventions: Behavioral: Shoulder Shaking
- Combined Verbal + Shoulder Tapping Group (Experimental)
  Interventions: Behavioral: Verbal Stimulation; Behavioral: Shoulder Tapping
- Combined Verbal + Shoulder Shaking Group (Experimental)
  Interventions: Behavioral: Verbal Stimulation; Behavioral: Shoulder Shaking

INTERVENTIONS:
Behavioral: Verbal Stimulation — Patients will wear headphones connected to a voice playback device that delivers pre-recorded verbal stimuli. Each voice message will last approximately 3 seconds, with a speech rate of 200-300 ms per character, and the volume will be set at a normal speaking level (60 dB). After each playback, there will be a 10-second interval before the next repetition, and the verbal stimulus will be played three times per intervention cycle.If the patient shows no eye opening or clear response, the standard verbal stimulation procedure will be repeated after a 3-minute interval, until a response is observed.
  Arms: Combined Verbal + Shoulder Shaking Group; Combined Verbal + Shoulder Tapping Group; Verbal Stimulation Group:
Behavioral: Shoulder Tapping — No audio will be played through the patient's headphones. Upon discontinuation of anesthetic agents, the investigator will begin tapping the patient's left shoulder. All operators will receive standardized training to ensure procedural consistency. The tapping frequency will be 2 taps per second, i.e., six taps within 3 seconds, paced using a metronome to maintain rhythm uniformity. Each tapping event (six taps over 3 seconds) will last 3 seconds, followed by a 10-second interval before the next tapping event.
  Arms: Combined Verbal + Shoulder Tapping Group; Shoulder Tapping Group
Behavioral: Shoulder Shaking — No audio will be played through the patient's headphones. Upon discontinuation of anesthetic agents, the investigator will begin gently shaking the patient's left shoulder.All investigators will undergo standardized training to ensure consistency of operation. Each shaking event (three shakes within 3 seconds) will last 3 seconds, followed by a 10-second interval before the next shaking event. Each intervention cycle will include three shaking events.
  Arms: Combined Verbal + Shoulder Shaking Group; Shoulder Shaking Group

SUMMARY:
This study intends to employ verbal stimulation, tactile stimulation, and kinetic stimulation as interventions during the emergence phase from general anesthesia to facilitate recovery.

DETAILED DESCRIPTION:
General anesthesia is an indispensable component of modern surgical practice. While its induction mechanisms have been relatively well elucidated, the mechanisms underlying emergence-namely the restoration of consciousness following anesthesia-remain incompletely understood. Emergence from anesthesia represents a critical stage of anesthetic management, with its efficiency and quality directly influencing postoperative recovery, patient safety, and the incidence of complications. Traditionally, anesthesia induction and emergence were considered to be symmetrical and passive processes, with emergence regarded as the reverse of induction that naturally occurs as anesthetic drug concentrations decline. However, recent advances in neuroscience suggest that anesthetic emergence is not merely a passive reversal but rather an actively regulated, multidimensional neurophysiological process with modulatory potential, and it is not entirely symmetrical to induction. Studies have demonstrated that neuronal activity in the cortex, activation patterns of brain regions, and neurotransmitter regulation during emergence differ substantially from those observed during induction. Key regulatory pathways implicated in this process include orexinergic neurons and the locus coeruleus-noradrenergic system. These findings provide a theoretical foundation for strategies aimed at facilitating emergence from general anesthesia.

Evidence further indicates that the sequence of functional recovery across different brain regions is heterogeneous during emergence. Clinical observations suggest that auditory perception is among the earliest sensory modalities to recover during anesthetic emergence. This phenomenon is of notable clinical significance, as it underlies the longstanding use of auditory interventions-such as calling a patient's name or giving verbal commands-in the operating room. Compared with other sensory modalities such as vision or nociception, auditory pathways regain responsiveness earlier. Although the precise neural mechanisms remain unclear, they are likely related to the auditory system, language processing circuits, and higher-order cortical integration of language. Recent advances in neuroimaging techniques, including electroencephalography (EEG) and functional magnetic resonance imaging (fMRI), provide further support for this perspective. For example, a previous study demonstrated via intracranial recordings that during propofol anesthesia, the core auditory cortex continued to generate early auditory evoked potentials and frequency-following responses to 50 Hz sound stimuli, indicating preserved early cortical responses. Similarly, another study showed that following loss of consciousness, the primary auditory cortex retained rapid responses to auditory input, whereas higher-order cortical responses were markedly attenuated. These findings suggest that auditory cortices can respond to external auditory stimuli even in the early stages of emergence when anesthetic concentrations remain pharmacologically significant, thereby supporting the use of auditory stimulation in facilitating recovery. Moreover, recent studies have investigated how specific linguistic content (e.g., a patient's own name) and acoustic characteristics (e.g., familiar voices) influence emergence quality. One study found that calling a patient's name elicited stronger responses and facilitated awakening more effectively than generic verbal cues. Similarly, another research reported that playback of maternal voice recordings shortened extubation time and reduced the incidence of emergence delirium in pediatric patients.

In addition to auditory stimulation, non-verbal somatosensory interventions are also commonly applied in clinical practice to promote emergence. Nevertheless, research on the role of such non-verbal stimulation in emergence from general anesthesia remains limited. Previous research demonstrated that acupuncture at acupoints such as Renzhong and Yongquan could accelerate the recovery of consciousness after general anesthesia. However, standardized protocols and robust evidence supporting the use of mechanical somatosensory stimulation to facilitate emergence are currently lacking. And its specific stimulation methods, intensity, timing of intervention, and safety parameters remain unclear.

Animal studies demonstrated in that electrical stimulation of glutamatergic neurons in the brainstem parabrachial nucleus can induce recovery of the righting reflex and behavioral arousal in mice under sustained isoflurane anesthesia, accompanied by a marked reduction in electroencephalographic δ waves. Subsequent studies further confirmed that stimulating glutamatergic neurons in the parabrachial nucleus accelerated anesthetic emergence, underscoring the critical role of this brainstem pathway in arousal regulation. The parabrachial nucleus is an important node in the central arousal network; its activation drives norepinephrine and dopamine release from the hypothalamus and brainstem, thereby enhancing cortical arousal. These findings suggest that peripheral somatosensory stimulation may ascend via spinal pathways to brainstem structures, thereby activating ascending arousal centers and accelerating recovery of consciousness. This provides a neurobiological basis for the use of peripheral somatosensory or spinal stimulation as non-invasive awakening strategies; however, clinical trials systematically validating such interventions remain lacking.

Although numerous studies have explored pharmacologic and non-pharmacologic approaches to accelerate emergence from general anesthesia, there is a paucity of randomized controlled trials evaluating the effectiveness and safety of non-verbal somatosensory stimulation. This approach is simple to implement, has a favorable safety profile, and does not increase healthcare costs. Its effects on emergence efficiency, emergence quality, and postoperative complications (e.g., delayed emergence, agitation) warrant systematic investigation, and such findings would provide evidence for clinical guidelines on anesthetic emergence.

Furthermore, electroencephalography (EEG), as a non-invasive method for real-time monitoring of brain function, is widely applied in assessing anesthetic depth and recovery of consciousness. Studies have shown that during emergence from general anesthesia, EEG exhibits characteristic changes, such as a reduction in high-amplitude slow waves, reappearance of α oscillations, and a gradual increase in β activity. Incorporating EEG frequency dynamics into the study design may help elucidate the neural mechanisms by which stimulation interventions modulate the arousal process, offering more direct neurophysiological evidence to optimize both monitoring and intervention strategies during anesthetic emergence.

In summary, the investigators propose to conduct a prospective, randomized controlled clinical trial to systematically investigate, in patients undergoing laparoscopic abdominal surgery under combined intravenous and inhalational general anesthesia, the effects of non-verbal somatosensory stimulation, either alone or in combination with verbal stimulation, compared with the conventional approach of verbal name-calling. Outcomes of interest include postoperative emergence time, quality, and safety. This study aims to provide robust scientific evidence to inform optimized intervention strategies for anesthetic emergence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 to 65 years, with American Society of Anesthesiologists (ASA) physical status I-III;
2. Scheduled for laparoscopic abdominal surgery, including gastric, colorectal, or biliary procedures;

Exclusion Criteria:

1. ASA physical status IV;
2. Body mass index (BMI) greater than 30 kg/m²;
3. Presence of underlying neurological dysfunction, cognitive impairment, or auditory disorders;
4. Neurological, cardiovascular, hepatic, or renal dysfunction;
5. Current use of antipsychotic medications or a history of psychiatric illness;
6. History of alcohol abuse or substance dependence;
7. Exposure to general anesthesia or sedation within 1 month prior to surgery;
8. Presence of intracranial implants or a history of epilepsy;
9. Known allergy to any drugs used in this study;
10. Preoperative use of electronic hearing aids or implanted auditory devices;
11. Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2025-10-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to first eye opening | Perioperative
  defined as the interval from discontinuation of anesthetic agents to the moment the patient opens both eyes in response to a verbal command and is able to keep them open for at least 5 seconds.

SECONDARY OUTCOMES:
Changes in EEG power | Perioperative
  Alterations in power across specific EEG frequency bands (e.g., Delta, Theta, Alpha, Beta) at the time of first eye opening
Time to target BIS values | Perioperative
  Time required for the BIS to reach 70, 80, and 90 after discontinuation of desflurane
Extubation time | Perioperative
  Interval from discontinuation of desflurane to removal of the endotracheal tube
Emergence agitation | Perioperative
  Highest score on the Riker Sedation-Agitation Scale (SAS) observed during emergence.
  The SAS ranges from 1 to 7, with higher scores indicating greater agitation and a worse outcome.
  Assessed from extubation to time before arrival in the post-anesthesia care unit.
Sedation depth after extubation | Perioperative
  Sedation level assessed using the Richmond Agitation-Sedation Scale (RASS) during emergence from anesthesia.
  The RASS ranges from -5 (unarousable) to +4 (combative), with higher scores indicating more agitation and lower scores indicating deeper sedation.
  Assessed from extubation to 30 minutes after arrival in the post-anesthesia care unit.
Hemodynamic parameters | Perioperative
  Mean arterial pressure (MAP) and heart rate (HR) recorded
Length of stay in PACU | Perioperative
  Length of stay in PACU
Postoperative analgesic use | Perioperative
  Total amount of analgesic administered in the PACU
Use of antiemetics | Perioperative
  Antiemetic medications administered in the PACU
Incidence of agitation in the PACU | Perioperative
  Proportion of patients with a Riker Sedation-Agitation Scale score ≥ 5. Assessed in the first 30 minutes after arrival in the post-anesthesia care unit.
Pain scores in the PACU | Perioperative
  Pain intensity assessed using the Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst possible pain.
  Higher scores indicate more severe pain. Assessed at 10 minutes, 20 minutes, and 30 minutes after arrival in the post-anesthesia care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available upon reasonable request from the corresponding author after publication and ethical approval. Data will be shared via email request to the corresponding author within 6 months after publication.

REFERENCES:
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Background] Rosow C, Manberg PJ. Bispectral index monitoring. Anesthesiol Clin North Am. 2001 Dec;19(4):947-66, xi. doi: 10.1016/s0889-8537(01)80018-3. PMID 11778388
- [Background] Cooper RM, O'Sullivan E, Popat M, Behringer E, Hagberg CA. Difficult Airway Society guidelines for the management of tracheal extubation. Anaesthesia. 2013 Feb;68(2):217. doi: 10.1111/anae.12139. No abstract available. PMID 23298360
- [Background] Jee D, Park SY. Lidocaine sprayed down the endotracheal tube attenuates the airway-circulatory reflexes by local anesthesia during emergence and extubation. Anesth Analg. 2003 Jan;96(1):293-7, table of contents. doi: 10.1097/00000539-200301000-00058. PMID 12505969
- [Background] Lee S, Sohn JY, Hwang IE, Lee HJ, Yoon S, Bahk JH, Kim BR. Effect of a repeated verbal reminder of orientation on emergence agitation after general anaesthesia for minimally invasive abdominal surgery: a randomised controlled trial. Br J Anaesth. 2023 Apr;130(4):439-445. doi: 10.1016/j.bja.2022.12.009. Epub 2023 Jan 23. PMID 36697272
- [Background] Hughes SW, Crunelli V. Thalamic mechanisms of EEG alpha rhythms and their pathological implications. Neuroscientist. 2005 Aug;11(4):357-72. doi: 10.1177/1073858405277450. PMID 16061522
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Lipp M, Schneider G, Kreuzer M, Pilge S. Substance-dependent EEG during recovery from anesthesia and optimization of monitoring. J Clin Monit Comput. 2024 Jun;38(3):603-612. doi: 10.1007/s10877-023-01103-4. Epub 2023 Dec 18. PMID 38108943
- [Background] Moody OA, Zhang ER, Vincent KF, Kato R, Melonakos ED, Nehs CJ, Solt K. The Neural Circuits Underlying General Anesthesia and Sleep. Anesth Analg. 2021 May 1;132(5):1254-1264. doi: 10.1213/ANE.0000000000005361. PMID 33857967
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Kreuer S, Biedler A, Larsen R, Altmann S, Wilhelm W. Narcotrend monitoring allows faster emergence and a reduction of drug consumption in propofol-remifentanil anesthesia. Anesthesiology. 2003 Jul;99(1):34-41. doi: 10.1097/00000542-200307000-00009. PMID 12826839
- [Background] Song D, White PF. Remifentanil as an adjuvant during desflurane anesthesia facilitates early recovery after ambulatory surgery. J Clin Anesth. 1999 Aug;11(5):364-7. doi: 10.1016/s0952-8180(99)00061-6. PMID 10526805
- [Background] Wang TX, Xiong B, Xu W, Wei HH, Qu WM, Hong ZY, Huang ZL. Activation of Parabrachial Nucleus Glutamatergic Neurons Accelerates Reanimation from Sevoflurane Anesthesia in Mice. Anesthesiology. 2019 Jan;130(1):106-118. doi: 10.1097/ALN.0000000000002475. PMID 30325744
- [Background] Muindi F, Kenny JD, Taylor NE, Solt K, Wilson MA, Brown EN, Van Dort CJ. Electrical stimulation of the parabrachial nucleus induces reanimation from isoflurane general anesthesia. Behav Brain Res. 2016 Jun 1;306:20-5. doi: 10.1016/j.bbr.2016.03.021. Epub 2016 Mar 10. PMID 26971629
- [Background] Gemma M, Nicelli E, Gioia L, Moizo E, Beretta L, Calvi MR. Acupuncture accelerates recovery after general anesthesia: a prospective randomized controlled trial. J Integr Med. 2015 Mar;13(2):99-104. doi: 10.1016/S2095-4964(15)60159-5. PMID 25797640
- [Background] Cao X, Wang B, Liu M, Li J. Effect of recorded mother's voice on emergence delirium in pediatric patients: a systematic review with meta-analysis. J Pediatr (Rio J). 2024 May-Jun;100(3):231-241. doi: 10.1016/j.jped.2023.08.008. Epub 2023 Oct 14. PMID 37844877
- [Background] Jung YS, Paik H, Min SH, Choo H, Seo M, Bahk JH, Seo JH. Calling the patient's own name facilitates recovery from general anaesthesia: a randomised double-blind trial. Anaesthesia. 2017 Feb;72(2):197-203. doi: 10.1111/anae.13688. Epub 2016 Oct 27. PMID 27786358
- [Background] Krom AJ, Marmelshtein A, Gelbard-Sagiv H, Tankus A, Hayat H, Hayat D, Matot I, Strauss I, Fahoum F, Soehle M, Bostrom J, Mormann F, Fried I, Nir Y. Anesthesia-induced loss of consciousness disrupts auditory responses beyond primary cortex. Proc Natl Acad Sci U S A. 2020 May 26;117(21):11770-11780. doi: 10.1073/pnas.1917251117. Epub 2020 May 12. PMID 32398367
- [Background] Nourski KV, Banks MI, Steinschneider M, Rhone AE, Kawasaki H, Mueller RN, Todd MM, Howard MA 3rd. Electrocorticographic delineation of human auditory cortical fields based on effects of propofol anesthesia. Neuroimage. 2017 May 15;152:78-93. doi: 10.1016/j.neuroimage.2017.02.061. Epub 2017 Feb 27. PMID 28254512
- [Background] Bonhomme V, Boveroux P, Brichant JF, Laureys S, Boly M. Neural correlates of consciousness during general anesthesia using functional magnetic resonance imaging (fMRI). Arch Ital Biol. 2012 Jun-Sep;150(2-3):155-63. doi: 10.4449/aib.v150i2.1242. PMID 23165875
- [Background] Zion-Golumbic E, Schroeder CE. Attention modulates 'speech-tracking' at a cocktail party. Trends Cogn Sci. 2012 Jul;16(7):363-4. doi: 10.1016/j.tics.2012.05.004. Epub 2012 May 30. PMID 22651956
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Mashour GA, Palanca BJ, Basner M, Li D, Wang W, Blain-Moraes S, Lin N, Maier K, Muench M, Tarnal V, Vanini G, Ochroch EA, Hogg R, Schwartz M, Maybrier H, Hardie R, Janke E, Golmirzaie G, Picton P, McKinstry-Wu AR, Avidan MS, Kelz MB. Recovery of consciousness and cognition after general anesthesia in humans. Elife. 2021 May 10;10:e59525. doi: 10.7554/eLife.59525. PMID 33970101
- [Background] Song XJ, Hu JJ. Neurobiological basis of emergence from anesthesia. Trends Neurosci. 2024 May;47(5):355-366. doi: 10.1016/j.tins.2024.02.006. Epub 2024 Mar 14. PMID 38490858
- [Background] Patel SR, Ballesteros JJ, Ahmed OJ, Huang P, Briscoe J, Eskandar EN, Ishizawa Y. Dynamics of recovery from anaesthesia-induced unconsciousness across primate neocortex. Brain. 2020 Mar 1;143(3):833-843. doi: 10.1093/brain/awaa017. PMID 32049333
- [Background] Zhang D, Wei Y. Distinct Neural Mechanisms Between Anesthesia Induction and Emergence: A Narrative Review. Anesth Analg. 2025 Jul 1;141(1):162-171. doi: 10.1213/ANE.0000000000007114. Epub 2024 Jun 11. PMID 38861419